CLINICAL TRIAL: NCT05682300
Title: "Incidence and Etiology of Complications Associated With Regional Anesthesia of Peripheral Nerves: a Prospective Study"
Brief Title: Incidence and Etiology of Complications Associated With Peripheral Nerves Blocks
Acronym: CARE
Status: Completed | Type: Observational
Sponsor: Hospital del Rio Hortega (Other)
Responsible Party: Principal Investigator, María Teresa Fernandez, Fernandez,Maria Teresa, MD, Principal investigator, Hospital del Rio Hortega
Other Study IDs: 22-EO069
Record Dates: First submitted 2022-12-19; First posted 2023-01-12 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Complication of Anesthesia
Keywords: peripheral nerve; regional anesthesia; complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient under regional anesthesia: patients who recieve peripheral nerve blocks as analgesic technique
  Interventions: Procedure: peripheral nerve block

INTERVENTIONS:
Procedure: peripheral nerve block — After signing the informed consent by the patient, specific for this observational study, the peripheral regional anesthesia technique will be performed following the usual practice of the anesthesiologist responsible for the surgery. Under standard monitoring and taking into account the necessary aseptic measures, either peripheral nerve blocks (for surgeries involving extremities) or fascial blocks (for surgeries involving the chest wall, abdomen, or spine) will be performed.

SUMMARY:
Procedures performed under regional anesthesia, especially peripheral nerve blocks (PNB) have increased markedly in recent decades. However, like any technical procedure, these techniques carry an implicit risk of complications.

The main objective of the study is to determine the incidence of complications associated with peripheral nerve blocks and fascial blocks in Spain.

DETAILED DESCRIPTION:
Introduction. The number of procedures performed under regional anesthesia, especially peripheral nerve blocks (BNP) have increased notably in recent decades due to the improvement in pain control and the quality of post-anesthetic recovery that they provide. However, like any technical procedure, these techniques carry an implicit risk of complications.

Purpose. The main objective of the study is to determine the incidence of complications associated with peripheral nerve blocks and fascial blocks in Spain.

Material and methods. The postoperative results regarding the complications of regional anesthesia of peripheral nerves will be evaluated in a national audit of a prospective observational cohort in which hospitals at the state level in which these regional techniques are routinely performed will participate. A minimum sample size has been calculated on a population of 100,000 patients and a 95% confidence interval of 1,390, assuming a complication rate of 0.2% based on previous publications.

Inclusion criteria correspond to patients older than 18 years scheduled for surgery with a peripheral regional anesthesia technique as the basis of anesthesia or as part of a multimodal analgesic strategy.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* ASA I- IV
* Being scheduled for surgery with peripheral and/or fascial nerve blocks as the basis of anesthesia or as part of a multimodal analgesic strategy.

Exclusion Criteria:

* Refusal of the patient to participate in the study
* Contraindication for performing the regional technique (People with infections in the area of the skin where the puncture must be performed, allergy to anesthetics, severe blood coagulation disorders, previous nerve damage).
* Motor or sensory deficit prior to surgery in the metameric area susceptible to performing the block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be carried out in all those hospitals nationwide that agree to be part of it.
  Each participating center will recruit patients for one year or until the estimated sample size is achieved.
  After signing the informed consent by the patient, specific to this observational study, the peripheral regional anesthesia technique will be performed following the usual practice of the anesthesiologist responsible for the surgery. Under standard monitoring and taking into account the necessary aseptic measures, either peripheral nerve blocks (for surgeries involving extremities) or fascial blocks (for surgeries involving the chest wall, abdomen, or spine) will be performed.
Sampling Method: Non-Probability Sample
Enrollment: 1390 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
rate of complications of peripheral nerve blocks | 2 years
  The main objective of the study is to determine the incidence of complications associated with peripheral nerve blocks and fascial blocks in Spain

SECONDARY OUTCOMES:
Etiology | 2 years
  Explain the etiology and mechanisms that contribute to nerve damage secondary to peripheral nerve blocks.
Number of Factors related | 2 years
  Explain the factors related to complications associated with fascial blocks.

CONTACTS AND LOCATIONS:
Overall Officials: María T Fernandez, Study Chair — Hospital del Rio Hortega
Locations (1):
- Judith Andres, Valladolid, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The study will be carried out in all those hospitals nationwide that agree to be part of it.
  Each participating center will recruit patients for one year or until the estimated sample size is achieved.